CLINICAL TRIAL: NCT05203757
Title: Weight-Bearing Cone Beam CT Arthrogram of the Ankle: a Lower Radiation Dose Technique to Evaluate Osteo-chondral Lesions or Cartilage Lesions: Is it the Future of the arthroCT?
Brief Title: Cone Beam CT (CBCT) Arthrogram of the Ankle in Assessement of Osteochondral or Cartilage Lesions
Acronym: Arthro-CBCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: APHP211118; 021-A01771-40 (Registry Identifier: IDRCB)
Record Dates: First submitted 2021-12-09; First posted 2022-01-24 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-04

CONDITIONS: Cartilage Lesion; Osteochondral Lesion
Keywords: Cartilage Lesion; Osteochondral Lesion; Osteochondral Defect; Cone Beam arthrogram; CBCT arthrogram; CT arthrogram; Weight bearing CBCT; Ankle

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Conventional CT-arthrogram + CBCT arthrogram (Experimental): Conventional CT-arthrogram + CBCT arthrogram (CBCT in the minutes following the conventional CT arthrogram).
  Routine care (arthroCT) and CBCT of ankle.
  Interventions: Procedure: ArthroCT scan; Procedure: CBCT

INTERVENTIONS:
Procedure: ArthroCT scan — Conventional CT arthrogram as routine care
Procedure: CBCT — Cone Beam CT scan.

SUMMARY:
This study aims to compare weight-bearing Cone Beam CT arthrogram and conventional CT arthrogram in assessement of patients with ankle osteo-chondral or cartilage lesions.

DETAILED DESCRIPTION:
Weight-bearing Cone Beam CT (CBCT) arthrogram, a technique with less radiation dose than conventional CT, is hypothesized non-inferior to conventional CT arthrogram to diagnose osteo-chondral (OCL) or cartilage lesions of the ankle.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥ 18 years;
* Patients require CT arthrogram of the ankle;
* Affiliated to a social security schema;
* Informed consent signed by patients.

Exclusion Criteria:

* Pregnant women;
* Impossibility of injection of intra-articular contrast product;
* Hypersensitivity reactions to iodinated contrast agent;
* Patient refusal;
* Patient under french AME scheme;
* Patient under guardianship by tutor or curator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2022-02-15 (Actual); Primary Completion 2023-08-15 (Actual); Study Completion 2023-08-15 (Actual)

PRIMARY OUTCOMES:
Localisation of the lesions | at baseline
  Localisation of cartilage and osteochondral lesions assessed by CT scan
Number of the lesions | at baseline
  Number of cartilage and osteochondral lesions assessed by CT scan
Size of the lesions | at baseline
  Size of cartilage and osteochondral lesions assessed by CT scan
Unstable displaced lesions | at baseline
  Displaced osteochondral fragment in the joint.
Unstable non-displaced lesions | at baseline
  Contrast enhanced fluid from the arthrogram surrounding the osteochondral fragment.

CONTACTS AND LOCATIONS:
Overall Officials: Mickael TORDJMAN, MD, Principal Investigator — Radiological department - Raymond Poincaré hospital - APHP
Locations (1):
- Radiological department, Raymond Poincaré hospital, APHP, Garches, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lopes R, Geffroy L, Padiolleau G, Ngbilo C, Baudrier N, Mainard D, Benoist J, Leiber Wackenheim F, Cordier G, Dubois Ferriere V, Freychet B, Barbier O, Amouyel T. Proposal of a new CT arthrographic classification system of osteochondral lesions of the talus. Orthop Traumatol Surg Res. 2021 Oct;107(6):102890. doi: 10.1016/j.otsr.2021.102890. Epub 2021 Mar 10. PMID 33713874
- [Background] Grunz JP, Pennig L, Fieber T, Gietzen CH, Heidenreich JF, Huflage H, Gruschwitz P, Kuhl PJ, Petritsch B, Kosmala A, Bley TA, Gassenmaier T. Twin robotic x-ray system in small bone and joint trauma: impact of cone-beam computed tomography on treatment decisions. Eur Radiol. 2021 Jun;31(6):3600-3609. doi: 10.1007/s00330-020-07563-5. Epub 2020 Dec 5. PMID 33280057
- [Background] Broos M, Berardo S, Dobbe JGG, Maas M, Streekstra GJ, Wellenberg RHH. Geometric 3D analyses of the foot and ankle using weight-bearing and non weight-bearing cone-beam CT images: The new standard? Eur J Radiol. 2021 May;138:109674. doi: 10.1016/j.ejrad.2021.109674. Epub 2021 Mar 20. PMID 33798932
- [Background] Posadzy M, Desimpel J, Vanhoenacker F. Staging of Osteochondral Lesions of the Talus: MRI and Cone Beam CT. J Belg Soc Radiol. 2017 Dec 16;101(Suppl 2):1. doi: 10.5334/jbr-btr.1377. PMID 30498800